CLINICAL TRIAL: NCT02404831
Title: An Evaluation of Web Based Pulmonary Rehabilitation- Pilot Study
Brief Title: An Evaluation of Web Based Pulmonary Rehabilitation
Acronym: webbasedPR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Research and Development (Other Government)
Responsible Party: Principal Investigator, Dr Lorna Paul, Dr, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L13099
Record Dates: First submitted 2014-12-02; First posted 2015-04-01 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Physiotherapy; Pulmonary Rehabilitation; Exercise; Telerehab
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional hospital-based PR (Active Comparator): Class based pulmonary rehabilitation
  Interventions: Other: Hospital-based PR
- Web-based PR (Experimental): web-based pulmonary rehab
  Interventions: Other: Web-based PR

INTERVENTIONS:
Other: Web-based PR — Participants will undertake web-based PR twice/week for 6 weeks in their own home. They will be given individual log-in details to access the website with access to exercises and education pages. Participants will be provided with a standardised exercise programme at the start of the study. The level of intensity of exercises will be progressed as appropriate on an individual basis for all participants in the group. Participant log-ins and diaries will be monitored remotely and participants will be telephone at weeks 2 and 4 by their physiotherapist to discuss their progress and, at this time, exercises may be progressed by changing the level of difficulty/intensity. This is done remotely by physiotherapy staff.
  Arms: Web-based PR
Other: Hospital-based PR — Participants allocated to this group will undertake hospital-based PR twice per week for 6 weeks in. Participants attend PR classes and complete a circuit based exercise class. The level of intensity of exercises will be progressed as appropriate on an individual basis for all participants in the group. Following each class they will receive educational information about their condition.
  Arms: Traditional hospital-based PR

SUMMARY:
The purpose of this pilot study is to compare a six week web-based pulmonary rehabilitation programme with traditional hospital-based pulmonary rehabilitation classes for people affected by COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a term used to describe a number of lung conditions characterised by irreversible damage to the airways causing airflow obstruction. Pulmonary Rehabilitation (PR) is a broad programme that helps improve the health and well-being of people with breathing difficulties, most commonly COPD. Participation in PR leads to improvements in exercise tolerance and functional ability, as well as a reducing breathlessness in everyday activities. It is traditionally an outpatient programme based in a hospital or community setting run by a multidisciplinary team, and usually lead by physiotherapy and nursing staff. Typically it includes a physical exercise programme, and advice and education on managing a chronic lung condition. The purpose of this pilot study is to compare a six week web-based pulmonary rehabilitation programme with traditional hospital-based pulmonary rehabilitation classes for people affected by COPD.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD
* Suitable for participation in the NHS Lanarkshire PR programme
* Independently mobile
* Access to the internet in their own home

Exclusion Criteria:

* Unstable cardiac or other health problems which may prevent participation in study
* Under the age of 18
* Pregnant
* Unable to read/understand English
* Unwilling to be randomised into PR delivered via the hospital or internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Shuttle Walk test at 6 weeks | 6 weeks
  analysis

SECONDARY OUTCOMES:
Change from baseline in Chronic Disease Questionnaire at 6 weeks | 6 weeks
  questionnaire

OTHER OUTCOMES:
Change from baseline in Hospital Anxiety and Depression Scale at 6 weeks | 6 weeks
Change from baseline in Borg Breathlessness Scale at 6 weeks | 6 weeks
Website evaluation questionnaire | 6 weeks
  questionnaire completed by Experimental Group only
Semi-structured telephone interviews | 6 weeks
  Qualitative interview conducted with Experimental Group only

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Paul, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Monklands Hospital, Airdrie, United Kingdom

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633